CLINICAL TRIAL: NCT00591864
Title: Comparison of Magnetic Resonance Imaging and Molecular Breast Imaging in Breast Diagnostic Evaluation
Brief Title: Comparison of MRI and Molecular Breast Imaging in Breast Diagnostic Evaluation
Acronym: MBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amy L. Conners, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 07-003397
Record Dates: First submitted 2007-12-21; First posted 2008-01-11 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: Benign breast disease; Breast; MRI; Mammography; Ultrasound; Molecular Breast Imaging; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Cystic Fibrosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Molecular Breast Imaging — Molecular breast Imaging is a new nuclear medicine technique for imaging the breast. It uses small filed of view semiconductor-based gamma cameras that use Cadmium Zinc Telluride detectors. These have superior spatial and energy resolution to conventional sodium iodide detectors.

SUMMARY:
The purpose of this study is to determine the sensitivity of Molecular Breast Imaging (MBI) relative to MRI of the breast in patients undergoing MRI for a clinical concern, or abnormal diagnostic mammogram and/or ultrasound study.

DETAILED DESCRIPTION:
Background: Breast MRI has excellent sensitivity, but is very expensive and suffers from low specificity. Additional benign biopsies are prompted by MRI in 24-40% of patients. Molecular Breast Imaging (MBI) is a new nuclear medicine technique developed at Mayo. Preliminary MBI results indicate a sensitivity of ~88% for the detection of tumors < 10 mm. The cost of an MBI procedure is expected to be a factor of 5 less than an MRI examination.

Hypothesis: MBI has a comparable sensitivity to MRI at a significantly lower cost.

Study Design: A total of 120 patients will be studied. All patients will have been scheduled for bilateral breast MRI at Mayo Clinic Rochester for a clinical concern, problem solving, or abnormal mammogram and/or ultrasound study. All patients will undergo MBI within 3 weeks of the MRI examination.

Potential Outcomes: This study will provide valuable information on the sensitivity of MBI relative to MRI, and to determine if this new technique can be eventually developed as an alternative to MRI for problem solving.

ELIGIBILITY:
Inclusion Criteria:

* This study will include a population of women aged 25 or older who are scheduled for a breast MRI examination at MAYO CLINIC ROCHESTER.
* Patients must not be lactating or pregnant.
* All women of child-bearing potential must have had a negative urine pregnancy test result within 2 days prior to the MBI study.
* women who are scheduled for a breast MRI examination for a clinical concern, problem solving or for further evaluation of invasive breast cancer (e.g. pre-operative staging of known breast cancer).

Exclusion Criteria:

* They are unable to understand and sign the consent form
* They are pregnant or lactating
* They are physically unable to sit upright and still for 40 minutes.
* The breast MRI is for screening purposes or to determine the status of breast augmentation.
* They have undergone breast surgery within the previous year

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic News Blog — http://newsblog.mayoclinic.org/2008/09/03/breast-cancer-molecular-breast-imaging-mammography/
- See also: Mayo Clinic You Tube Channel — http://www.youtube.com/watch?v=DOQBLe8MdH0

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Imaged With MBI and MRI: The group includes patients who underwent both MBI and breast MRI within the same 3 week period.
Period: Overall Study
Arm/Group | Participants Imaged With MBI and MRI
Started | 89
Completed | 84
Not Completed | 5
Not completed — Incomplete Imaging | 5

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: There are no arms or subgroups in this study.
Arm/Group | Study Participants
Number analyzed (Participants) | 89
Age, Continuous [Mean (Full Range); unit: Years] | 53 [35 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity on the Per Patient Level
Description: Sensitivity is the number of women with breast cancer detected per number of women with breast cancer diagnosed by surgery or biopsy.
Time Frame: within 1 week of surgery or biopsy
Population: In the 84 patients who completed the study 28 were diagnosed with breast cancer.
Measure: Number; unit: participants
Arm/Group | Study Participants
Number analyzed (Participants) | 28
participants
  Sensitivity by MBI | 25
  Sensitivity by MRI | 27

2. Secondary Outcome: Sensitivity on the Per Tumor Level
Description: Number of tumors detected per number of tumors diagnosed on surgery or biopsy.
Time Frame: within 1 week of surgery or biopsy
Measure: Number; unit: tumors
Units Other Than Participants: tumors
Arm/Group | Participants Imaged With MBI and MRI
Number analyzed (Participants) | 28
Number analyzed (tumors) | 37
tumors
  sensitivity by MBI | 32
  sensitivity by MRI | 36

3. Secondary Outcome: Specificity
Description: The number of women with negative imaging test per number of women without cancer.
Time Frame: at least one year following imaging
Measure: Number; unit: participants
Arm/Group | Participants Imaged With MBI and MRI
Number analyzed (Participants) | 56
participants
  specificity by MBI | 38
  specificity by MRI | 37

ADVERSE EVENTS:
Arm/Group | Study Participants
Serious Adverse Events (participants affected / at risk) | 0/89
Other Adverse Events (participants affected / at risk) | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes